CLINICAL TRIAL: NCT05644639
Title: StimRouter Genicular NeuromoduLation for Chronic KnEe OsteoArthritic Pain Management
Brief Title: Study of StimRouter for Chronic Knee OA Pain
Acronym: GLEAM
Status: Completed | Type: Observational
Sponsor: Bioventus LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PNS-22-01
Record Dates: First submitted 2022-11-16; First posted 2022-12-09 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis, Knee
Keywords: StimRouter; Osteoarthritis; Neuromodulation; Knee Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: StimRouter Neuromodulation System — The StimRouter device is indicated for pain management in adults who have severe, intractable chronic pain of peripheral nerve origin and as an adjunct to other modes of therapy (e.g., medications). The StimRouter device is not intended to treat pain of craniofacial nerve origin.
  Other Names: StimRouter

SUMMARY:
The goal of this study is to evaluate the use of StimRouter Neuromodulation System (StimRouter) in adult subjects with an established diagnosis of primary femorotibial osteoarthritis in the target knee (Kellgren-Lawrence ≥1) who have surgical contraindications to undergo a knee joint arthroplasty procedure. The main questions it aims to answer are:

1. To assess the effect of the StimRouter Neuromodulation System to manage joint pain in patients with symptomatic OA of the knee who are surgically contraindicated to undergo a knee joint arthroplasty
2. To assess the effect of StimRouter on joint stiffness, function and patient quality of life

Participants will have StimRouter leads implanted then clinic visits will be scheduled for follow-up at Week 2, Month 3 and Month 6 (End of Study (EOS) or Early Termination (ET)).

DETAILED DESCRIPTION:
This study will be a single-center, single-arm, open label pilot study evaluating the safety and efficacy of the StimRouter Neuromodulation System as a peripheral nerve stimulator targeting knee joint innervation of moderately to severely symptomatic subjects with OA of the knee who are non-eligible to undergo a joint arthroplasty at the target knee.

Up to 30 subjects will be enrolled and participate in the study. Clinic visits will be scheduled at Screening, Stimulation Trial Procedure, Trial Assessment Visit, Implant Procedure and Follow-up Week 2, Month 3 and Month 6 (End of Study (EOS) or Early Termination (ET)).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 21 years of age at the time of giving informed consent
2. Radiographic disease Stage ≥ 1 in the target knee according to the Kellgren-Lawrence grading of knee OA
3. Knee joint arthroplasty procedure is contraindicated
4. Full understanding of the requirements of the study and willingness to comply with all study visits and assessments
5. Subjects must have read and understood the informed consent form, and must have signed it prior to any study-related procedure being performed

Exclusion Criteria:

1. Subject has undergone previous joint arthroplasty procedure (partial, total, patella-femoral) to the index knee
2. Unresolved effusion of the target knee clinically requiring aspiration within 12 weeks prior to Visit 1 (Baseline)
3. Treatment of the index knee with systemic or intra-articular corticosteroids (e.g., methylprednisolone) within 6 weeks prior to Visit 1 (Baseline)
4. Visco-supplementation (e.g., hyaluronic acid) in the index knee within 6 weeks prior to Visit 1 (Baseline)
5. Subject has an active systemic infection or an active local infection in or near the index knee joint, or has a previous history of joint infection.
6. Subject with bleeding disorders or active anticoagulation that cannot be stopped for a few days prior to the time of the surgical procedure.
7. Subject who has an active or existing skin disorder or irritation, which, in the opinion of the Investigator, precludes the use of skin gel electrodes.
8. Subjects has or plans to have a pacemaker, defibrillator, cochlear implant, and/or a sleep apnea implant.
9. Subject has or plans to have a Spinal Cord Stimulator (SCS), Peripheral Nerve field Stimulation system (PNfS), Dorsal Root Ganglion system (DRG), or implantable infusion pump.
10. Subject who currently requires or is likely to require Magnetic Resonance Imaging (MRI) within the MRI exclusion zone: the entire PNS lead must be at least 50 cm from the center of the MRI system's bore (the iso-center) and at least 16 cm outside of the MRI coil measured from the edge of the MRI coil.
11. Female subject who is pregnant or nursing or plans to become pregnant during the study. The effects of electrical stimulation on pregnancy are not known. Do not use electrical stimulation (including StimRouter) during pregnancy.
12. Any condition and findings in the medical history or in the pre-study assessments, that in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
13. Comorbid conditions that could affect pain assessment of the target knee, including, but not limited to, inflammatory rheumatic conditions such as rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subjects with an established diagnosis of primary femorotibial OA in the target knee (Kellgren-Lawrence ≥1) who have surgical contraindications to undergo a knee joint arthroplasty procedure
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Knee Pain | The primary endpoint is at Month 3 post permanent implantation.
  Change in pain with a Numeric Rating Scale (minimum 0 and maximum 10) from Baseline to 3 months after treatment
Knee Pain | The primary endpoint is at Month 3 post permanent implantation.
  Change in pain from Baseline to Month 3 in knee health as assessed by the KOOS-12 questionnaire. The KOOS-12 questionnaire is a 12-item measure derived from the original 42 item Knee injury and Ostoearthritis Outcome Score (KOOS). KOOS-12 contains 4 KOOS Pain items, 4 KOOS Function (Activities of Daily Living and Sport/Recreation) items, and 4 KOOS Quality of Life (QOL) items.

SECONDARY OUTCOMES:
Serious Adverse Events (SAEs) | The primary endpoint is at Month 3 post permanent implantation.
  Frequency and proportion of device, or procedure-related Serious Adverse Events (SAEs) in subjects who receive permanent implant of the StimRouter Neuromodulation System
Serious Adverse Events (SAEs) | Patients will continue to be followed up to Month 6 to gather additional efficacy and safety data.
  Frequency and proportion of device, or procedure-related Serious Adverse Events (SAEs) in subjects who receive permanent implant of the StimRouter Neuromodulation System
Adverse Events (AEs) | The primary endpoint is at Month 3 post permanent implantation.
  Frequency and proportion of device, or procedure-related non-serious adverse events (AEs) in subjects who receive permanent implant of the StimRouter Neuromodulation System
Adverse Events (AEs) | Patients will continue to be followed up to Month 6 to gather additional efficacy and safety data.
  Frequency and proportion of device, or procedure-related non-serious adverse events (AEs) in subjects who receive permanent implant of the StimRouter Neuromodulation System
Secondary Interventions | The primary endpoint is at Month 3 post permanent implantation.
  Rate of secondary interventions (e.g. surgical or intra-articular injection) to the index knee
Secondary Interventions | Patients will continue to be followed up to Month 6 to gather additional efficacy and safety data.
  Rate of secondary interventions (e.g. surgical or intra-articular injection) to the index knee
Knee Pain | Patients will continue to be followed up to Month 6 to gather additional efficacy and safety data.
  Change in pain with a Numeric Rating Scale (minimum 0 and maximum 10) from Baseline to 6 months after treatment
Knee Health | Patients will continue to be followed up to Month 6 to gather additional efficacy and safety data.
  Change in pain from Baseline to Month 6 in knee health as assessed by the KOOS-12 questionnaire. The KOOS-12 questionnaire is a 12-item measure derived from the original 42 item Knee injury and Ostoearthritis Outcome Score (KOOS). KOOS-12 contains 4 KOOS Pain items, 4 KOOS Function (Activities of Daily Living and Sport/Recreation) items, and 4 KOOS Quality of Life (QOL) items.
Pain Experience | The primary endpoint is at Month 3 post permanent implantation.
  the change from baseline to Month 3 in pain experience (pain catastrophizing) as assessed by the PCS questionnaire scale score.
Pain Experience | Patients will continue to be followed up to Month 6 to gather additional efficacy and safety data.
  the change from baseline to Month 6 in pain experience (pain catastrophizing) as assessed by the PCS questionnaire scale score
Treatment Satisfaction Scores | Patients will continue to be followed up to Month 6 to gather additional efficacy and safety data.
  Treatment Satisfaction is measured using a 5 question questionnaire with answers ranging from "Very Satisfied" to "Very Dissatisfied"
Forgotten Joint Score (FJS) | The primary endpoint is at Month 3 post permanent implantation.
  The FJS-12 Questionnaire comprises measures for assessment of joint-specific patient reported outcomes that focuses on subject's awareness of affected joint in everyday life. Joint awareness defined as any unintended perception of a joint. Subjects rate awareness of their knee joint in 12 questions with a 5-point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". Scores are summed & linearly transformed in a 0-100 scale with a high value reflecting subject's ability to forget the affected knee joint during daily living activities.
Forgotten Joint Score (FJS) | Patients will continue to be followed up to Month 6 to gather additional efficacy and safety data.
  The FJS-12 Questionnaire comprises measures for assessment of joint-specific patient reported outcomes that focuses on subject's awareness of affected joint in everyday life. Joint awareness defined as any unintended perception of a joint. Subjects rate awareness of their knee joint in 12 questions with a 5-point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". Scores are summed & linearly transformed in a 0-100 scale with a high value reflecting subject's ability to forget the affected knee joint during daily living activities.
Health-Related Quality of Life (HRQOL) | The primary endpoint is at Month 3 post permanent implantation.
  the change from baseline to Month 3 in Health-Related Quality of Life (HRQOL) as assessed by the PROMIS-10 Global Health questionnaire. The PROMIS-10 is a 10 question questionnaire with answers ranging from "Excellent" to "Poor"
Health-Related Quality of Life (HRQOL) | Patients will continue to be followed up to Month 6 to gather additional efficacy and safety data.
  the change from baseline to Month 6 in Health-Related Quality of Life (HRQOL) as assessed by the PROMIS-10 Global Health questionnaire. The PROMIS-10 is a 10 question questionnaire with answers ranging from "Excellent" to "Poor"
Treatment Satisfaction Scores | The primary endpoint is at Month 3 post permanent implantation.
  Treatment Satisfaction is measured using a 5 question questionnaire with answers ranging from "Very Satisfied" to "Very Dissatisfied"
Treatment Expectation Scores | The primary endpoint is at Month 3 post permanent implantation.
  Treatment Expectation is measured using a 3 question questionnaire with subjects assessing their expectations of treatment ranging from "Too Low - I'm a lot better than I thought" to "Too High - I'm somewhat worse than I thought"
Treatment Expectation Scores | Patients will continue to be followed up to Month 6 to gather additional efficacy and safety data.
  Treatment Expectation is measured using a 3 question questionnaire with subjects assessing their expectations of treatment ranging from "Too Low - I'm a lot better than I thought" to "Too High - I'm somewhat worse than I thought"

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Mendelson, MD, Principal Investigator — Mendelson Kornblum Orthopedics
Locations (1):
- Mendelson Kornblum Orthopedic and Spine Specialists, Livonia, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided